CLINICAL TRIAL: NCT06353490
Title: The Clinical Performance Validation of Electronic Thermometer and Infrared Thermometers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Geon-111001
Record Dates: First submitted 2024-03-20; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Febrile; Healthy
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects: 0 up to 1 year (Other): Collecting temperatures using the "Geon" Digital, Infrared Ear and Infrared Forehead thermometer
  Interventions: Device: Infrared Forehead Thermometer (GE-TF03); Device: Infrared Ear Thermometer (GE-TE06); Device: Electronic Thermometer (MT-B321FB); Device: Electronic Thermometer (MT-B231)
- Subjects: Older than 1 year and younger than 5 years (Other): Collecting temperatures using the "Geon" Digital, Infrared Ear and Infrared Forehead thermometer
  Interventions: Device: Infrared Forehead Thermometer (GE-TF03); Device: Infrared Ear Thermometer (GE-TE06); Device: Electronic Thermometer (MT-B321FB); Device: Electronic Thermometer (MT-B231)
- Subjects: Older than 5 years (Other): Collecting temperatures using the "Geon" Digital, Infrared Ear and Infrared Forehead thermometer
  Interventions: Device: Infrared Forehead Thermometer (GE-TF03); Device: Infrared Ear Thermometer (GE-TE06); Device: Electronic Thermometer (MT-B321FB); Device: Electronic Thermometer (MT-B231)

INTERVENTIONS:
Device: Infrared Forehead Thermometer (GE-TF03) — Infrared Forehead Thermometer (GE-TF03) is an investigational device intended to measure body temperature on the forehead. GE-TF03 took three measurements for each subject.
Device: Infrared Ear Thermometer (GE-TE06) — Infrared Ear Thermometer (GE-TE06) is an investigational device intended to measure body temperature in the ear canal. GE-TF06 took three measurements for each subject.
Device: Electronic Thermometer (MT-B321FB) — Electronic Thermometer (MT-B321FB) is an investigational device intended to measure body temperature on the temporal artery. MT-B321FB took three measurements for each subject.
Device: Electronic Thermometer (MT-B231) — Electronic Thermometer (MT-B231) is a reference device that measured axillary temperature one time for each subject.

SUMMARY:
Geon Corporation develops ear thermometers and forehead thermometers that use infrared measurement technology to measure human body temperature. This study verify the accuracy and repeatability of investigational devices. Efficacy verification is carried out by comparing with the referent medical devices.

The main objectives of this study are:

1. To verify that the investigational devices and the reference medical devices have a reasonable deviation value.
2. To verify the consistency of repeated measurements of investigational devices.

DETAILED DESCRIPTION:
This Study carried out in accordance with the ISO 80601-2-56: 2017, which included definitions for the age groups and sample sizes, the definition of fever, the flowchart for relevant procedures, and statistical methods for clinical performance.

All subjects were measured by the reference device (electronic thermometer MT-B231) and three investigational devices under test evaluation (infrared forehead thermometer GE-TF03, infrared ear thermometer GE-TE06, and electronic thermometer MT-B321FB). For each subject, the reference device measured one time and each investigational device measured three times respectively.

ELIGIBILITY:
Inclusion Criteria:

* Newborn to 80 years old adult
* Male or Female
* The subject or parent/guardian can talk to the researcher, understand the content of the study after researcher's explanation and agree to sign the subject's consent form, and is willing to accept the trial procedure.

Exclusion Criteria:

* Currently have signs or symptoms of infection or inflammation at the temperature measurement site (axillary, forehead, ear canal)
* The forehead cannot be fully exposed to the environment for more than 15 minutes
* Using cooling blankets, fans, or placing ice cubes on the forehead
* There is a catheter placed in the ear
* Use of antipyretics (such as aspirin, ibuprofen), barbiturates, antipsychotics in the past 2 hours
* Received thyroxine, corticosteroids or immunotherapy in the past 7 days
* Subject has been diagnosed with cognitive impairment or has a history of dementia, mental illness, mental illness, pervasive developmental disorder, illicit drug use or alcoholism, etc.
* Pregnant women
* The researcher considers that the subject is not suitable for participating in this trial, such as taking any drugs that may change body temperature
* Participated in clinical trials of investigational drugs within the last 30 days
* The subject is unwilling to sign the subject's consent form

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-08-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Bias | Through study completion, an average of 2 years
  Mean Difference between investigational thermometer and reference thermometer.
Limits of Agreement | Through study completion, an average of 2 years
  The magnitude of a potential disagreement between investigational thermometer and reference thermometer.
Clinical Repeatability | Through study completion, an average of 2 years
  Pooled standard deviation of triplicate measurements over the entire population of subject

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Te Lei, Principal Investigator — Hsinchu MacKay Memorial Hospital
Locations (2):
- Taiwan (2):
  - Hsinchu MacKay Memorial Hospital, Hsinchu
  - HsinChu Municipal MacKay Memorial Hospital, Hsinchu